CLINICAL TRIAL: NCT00685269
Title: The Safety and Efficacy of Eszopiclone in Subjects With Mild to Moderate Obstructive Sleep Apnea Syndrome
Brief Title: Safety and Efficacy of Eszopiclone With Mild to Moderate Obstructive Sleep Apnea Syndrome (OSAS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 190-028
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; OSAS
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): eszopiclone 3 mg QD
  Interventions: Drug: Eszopiclone
- B (Placebo Comparator): placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 3 mg QD
  Other Names: Lunesta; (S)-Zopliclone
  Arms: A
Drug: Placebo — Placebo tablet
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the hypnotic efficacy of ezopiclone in subjects with mild to moderate OSAS.

DETAILED DESCRIPTION:
Sleep apnea is a sleep disorder characterized by pauses in breathing during sleep. This study will compare the use of eszopiclone to placebo for subjects with mild to moderate obstructive sleep Apnea syndrome (OSAS). Frequency and duration of apnea and hypopnea episodes, oxygen saturation, objective sleep parameters and safety information will be collected in this study. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* The subject is capable of understanding and complying with the protocol and has signed the informed consent document, including the privacy authorization. Female subjects of childbearing potential must sign the Women of Childbearing Potential Addendum to the informed consent form.
* Male and female subjects between 35 and 64 years of age, inclusive, with mild to moderate obstructive sleep apnea syndrome (AHI range ≥10 and ≤40).
* Females considered not of childbearing potential must be surgically sterile or greater than one-year post menopausal, defined as a complete cessation of menstruation for at least one year.
* Subjects must use continuous positive airway pressure (CPAP).
* Subjects must be in general good health based on screening physical examination (defined as the absence of any clinically relevant abnormalities), medical history, 12-lead ECG, and clinical laboratory values (hematology, serum chemistry and urinalysis).

Exclusion Criteria:

* Subject has any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, respiratory, hepatic, or renal systems.
* Subject has a history of, or current malignancy except for non melanomatous skin cancer.
* Subject tests positive at screening for hepatitis B surface antigen or hepatitis C antibody, or the subject has a history of a positive result.
* Subject is known to be seropositive for human immunodeficiency virus (HIV).

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-08; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
AHI (frequency of apnea and hypopnea episodes). | Nights -14, 1, 2, 8, 9

SECONDARY OUTCOMES:
The mean duration of apnea and hypopnea episodes | Nights -14, 1, 2, 8, 9
Oxygen saturation during apnea and hypopnea | Nights -14, 1, 2, 8, 9
The number of arousals during apnea and hypopnea | Nights -14, 1, 2, 8, 9
Objective sleep parameters as measured by PSG (i.e., latency to persistent sleep, sleep efficiency, and wake time after sleep onset | Nights -14, 1, 2, 8, 9

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atlanta, Georgia
  - Cincinnati, Ohio